CLINICAL TRIAL: NCT07291427
Title: Safety and Efficacy of Chronic Subdural Hematoma Embolization With Detachable Coils
Brief Title: Chronic Subdural Hematoma Embolization With Detachable Coils
Acronym: SEED
Status: Not yet recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: John Muir Health (Other); Carondelet Neurological Institute (Unknown)
Responsible Party: Principal Investigator, Christopher P Kellner, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-25-01365
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Subdural Hemorrhage (cSDH)
Keywords: Subdural hemorrhage; Coils; Middle meningeal artery
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Hematoma, Subdural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Participants with cSDH: All participants enrolled will be treated with the Balt coils.
  1. MMA embolization: Utilize Balt Coils as stand-alone with or without other embolics treatment.
  2. MMA embolization: Utilize Balt Coils in combination with or without embolics in surgical or bedside evacuation, such as:
     1. MMA embolization in combination with Balt coils post-surgical debridement, or
     2. MMA embolization using Balt coils alone, pre- or post-surgical debridement.
  Interventions: Device: Balt coils: (Balt USA, LLC); Procedure: MMA embolization

INTERVENTIONS:
Device: Balt coils: (Balt USA, LLC) — MMA embolization utilizing Balt Coils
  Other Names: Optima; OptiMax; OptiBlock; Optima series line extensions
Procedure: MMA embolization — surgical or bedside evacuation
  pre or post-surgical debridement

SUMMARY:
This is a prospective, multi-center, post market registry study designed to evaluate the safety and efficacy of treatment with Balt coils in patients with chronic subdural hematoma (cSDH).

DETAILED DESCRIPTION:
The primary objective of this observational registry study is to assess the safety and efficacy of Balt Coils as an adjunct to middle meningeal artery (MMA) embolization in a real-world setting among patients undergoing treatment for chronic subdural hematoma (cSDH), and explore correlations between patient characteristics, clinical characteristics, and outcomes. By collecting comprehensive, real-world data, the registry will characterize procedural inputs, document clinical and radiographic outcomes, and explore variation in technique and practice setting. The overarching goal is to generate a more complete understanding of Middle Meningeal Artery Embolization (MMAE) in diverse clinical environments, inform future prospective studies, and guide evidence-based adoption of this evolving therapy. Patients may be treated with Balt coils regardless of enrollment in the study as the decision to place the coils should be made independently as per standard of care and prior to enrollment in the study.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18
* Patients experiencing unilateral or bilateral non-acute subdural hematoma confirmed by CT imaging. Acute on Chronic or mixed density hematoma allowed.
* A clinical decision has been made to use coiling and/or embolics as treatment, with or without surgical debridement, independently as per standard of care and prior to enrollment in the study.
* Signed informed consent obtained by patient or Legal Authorized Representative (LAR)

Exclusion criteria:

* Primary acute SDH
* Prior MMAE in target territory
* Premorbid mRS > 3
* Common carotid stenosis >70% or prior carotid stent placement
* Significant medical contraindication to angiography (kidney failure/disease)
* Anatomical variations that would make MMA embolization difficult or unsafe
* Currently participating in an investigational (drug, device, etc.) clinical trial that may confound study endpoints
* Pregnancy
* Life expectancy ≤ 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic chronic subdural hematoma (cSDH), with or without previous surgical evacuation that need additional treatment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in hematoma volume | 180 days
  Change in hematoma volume based on CT imaging
Change in maximal thickness | 180 days
  Change in maximal thickness based on CT imaging
Change in midline shift | 180 days
  Change in midline shift (mm) based on CT imaging
Number of periprocedural major disabling stroke or any death | 30 days
  Number of periprocedural major disabling stroke or any death
Number of participants with symptomatic recurrence progression requiring retreatment | 180 days
  Number of participants with symptomatic recurrence progression of the SDH requiring retreatment

SECONDARY OUTCOMES:
Number of Device-related adverse events (AE), serious adverse events (SAE), and procedural-related SAE | 180 days
  Number of Adverse events and serious adverse events related to the device as assessed by an independent medical monitor
Number of Acute successful embolization of the target vessel | Immediately post-procedure
  Determination of successful embolization based on angiographic imaging
Change in EuroQoL 5 dimensions 5 levels (EQ-5D-5L) | 180 days
  The EQ-5D is a generic instrument for describing and valuing health. The new version includes the 5 levels of severity in each of the existing five EQ-5D dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and now called the EQ-5D-5L, each assessed on a 5-point scale (1=no problem, 2=slight problems, 3=moderate problems, 4=severe problems, 5=extreme problems). Participants score each dimension based on their health that day and their responses are used to generate a health index score. Index scores could range from <0 (a health state equivalent to dead with negative values representing a state worse than dead) to 1 (full health). Lower scores indicate a higher QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kellner, Principal Investigator — Icahn School of Medicine at Mount Sinai; Benjamin Yim, Principal Investigator — John Muir Health; Alexander Coon, Principal Investigator — Carondelet Neurological Institute
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Upon the completion of the study, Mount Sinai's data management team will clean and analyze all data in preparation of manuscript writing and publication. Data that will be shared and published will be that of all participants combined to protect individual patient privacy and confidentiality.